CLINICAL TRIAL: NCT02220101
Title: Temperature Measurement in Surgical and Intensive Care Patients - Comparison of Four Measurement Methods
Acronym: Temp
Status: Completed | Type: Observational
Sponsor: Sykehuset i Vestfold HF (Other)
Collaborators: 3M (Industry)
Responsible Party: Principal Investigator, Espen Lindholm, Chief of Department of Anesthesiology section, Sykehuset i Vestfold HF
Other Study IDs: 1A
Record Dates: First submitted 2014-02-06; First posted 2014-08-19 (Estimated); Last update posted 2023-01-04 (Actual); Status verified 2023-01

CONDITIONS: Hypothermia; Hyperthermia
Keywords: hypothermia; core temperature; temperature measurement methods
MeSH Terms: conditions — Hypothermia; Hyperthermia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Comparison of four methods for measuring temperature perioperatively in patients scheduled for laparoscopic surgery and intensive care patients who are hypo-, normo-and hyper terme; Bladder Monitoring, Nasopharyngeal, SpotOn TM, Zero heat flux method and Temporal Scanner. The study is a single-center, observational study carried out by the Central Surgical and Intensive Section at Vestfold Hospital Trust.

DETAILED DESCRIPTION:
Issues

* Perioperative hypothermia is associated with several serious complications and therefore most likely to be avoided. Monitoring of body temperature is therefore required perioperatively .
* There are in the literature concerns that some methods of measuring temperature perioperatively is accurate enough and whether they reflect core temperature adequate.
* Some authors have questioned whether temporal scanner (TS ) - and nasopharynx ( NP) - measurements are accurate enough to measure the actual core temperature. Much of the research on TS measurements have been done on children and newborns in an intensive setting, but little perioperatively .

A total of 120 patients will be included ; 60 at Central Operations and 60 at Intensive Section at the Vestfold Hospital Trust. Duration of inclusion will be approximately one year . Starting around January 2014. The study emanates from Vestfold Hospital Trust and was designed by Espen Lindholm who is responsible for the project , Camilla B Norén who is principal investigator and project manager. Kjetil G Ringdal , Karl - André Wian and Knut Arvid Kirkebøen (University Hospital of Oslo ) are supervisors. The study is supported by research, Vestfold Hospital Trust and 3M Company Norway (study material ) and it is applied Regional Ethics Committee. Patients will not get different treatment than standard treatment in hospital and it causes no follow-up calls or hospital visits. All patients (if possible) give written consent for participation.

ELIGIBILITY:
Inclusion Criteria:

Surgical Patient group:

* > 18 years
* ASA 1-3
* Laparoscopic surgery
* Elective surgery

Intensive Patient group:

* > 18 years
* Defined as intensive patient
* ASA 1-5

Exclusion Criteria:

Surgical Patient group:

* BMI> 30 kg/m2
* No bladder (ileum-bladder)
* Known malignant hyperthermia
* Malformations of the face that prevents nasopharynx and temporal scanner measurements
* Patient is participating in another study that may influence the results of the Tempstudy
* The patient is not competent to give consent, eg severe dementia
* The patient INR> 2.0 and / or Trc <50

Intensive Patient group:

* BMI> 30 kg/m2
* No bladder (ileum-bladder)
* Malformations of the face that prevents nasopharynx and temporal scanner measurements
* Hypothermic patient below 32 ° C (bladder temperature)
* Hyperterm patient over 40 ° C (bladder temperature)
* Active cooling of the bladder
* The patient is under ongoing cooling or heating
* Patient is participating in another study that may influence the results of the Tempstudy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Laparoscopic surgery and in ICU patients
Sampling Method: Non-Probability Sample
Enrollment: 95 (Actual)
Dates: Start 2014-04; Primary Completion 2023-01 (Actual); Study Completion 2023-01 (Actual)

PRIMARY OUTCOMES:
Temperature difference measured with different measuring methods | Timepoints during surgery; Every 20th minute. In intensive patients: 3 measurements during 1 hour (every 20th minute)
  The difference in temperature between the temperature measured by the current reference method bladder temperature and the temperature measured with Temporal Scanner, SpotOn and nasopharynx through the entire operational sequence (from first to last measurement) and three individual measurements at 20 minute intervals of intensive care patients.

SECONDARY OUTCOMES:
Number of patients with 1) Sore after Sticker (SpotOn) 2) epistaxis during hospital stay as a measure of safety and tolerability. | Hospital discharge
  An average of 10 days

CONTACTS AND LOCATIONS:
Overall Officials: Espen Lindholm, M.D., Study Director — Departement of Anesthesiology, Vestfold Hospital Trust
Locations (1):
- Vestfold Hospital Trust, Tønsberg, Norway